CLINICAL TRIAL: NCT04803903
Title: Is The Hypotension Probability Indicator With Goal Directed Haemodynamic Treatment Useful In Predicting And Treating Hypotension In General Anesthesia Patients?
Brief Title: HPI Index With GDHT in Predicting Hypotension In General Anesthesia Patients
Status: Completed | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Tatiana Sidiropoulou, Associate Professor of Anesthesiology, Attikon Hospital
Other Study IDs: 11.15.2018
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Hypotension During Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HPI + GDHT treatment: HPI + GDHT treatment using the FlowTraQ sensor and EV1000 monitor with the HPI algorithm incorporated following our protocol for hemodynamic treatment (fluids, vasopressors and inotropes) administered
  Interventions: Device: Flotraq Sensor with EV1000 incorporating the HPI algorithm
- Control: Conventional treatment with invasive blood pressure monitoring. Administration of fluids and/or vasopressors are guided by standard hemodynamic parameters at the discretion of the attending physician.

INTERVENTIONS:
Device: Flotraq Sensor with EV1000 incorporating the HPI algorithm — The HPI algorithm is only available on the EV1000, Hemosphere and Flotrac monitoring systems and requires the use of a Flotrac sensor connected to an arterial line (Edwards Lifesciences Corp., Irvine, CA, USA). The Flotrac sensor has a splitter which enables the splitting of the arterial blood pressure signal to facilitate a blood pressure signal on both the anesthesia machine monitor (standard care) and the HemoSphere monitor (study).
  In the intervention arm we asked the anesthesiologist and anesthesia nurse to use the study treatment flowchart . If the HPI alarm goes off, which entails both a sound and a flickering light, we ask the anesthesiologist to act upon this alarm immedietaly. Use of the study treatment flowchart ensures that the anesthesiologist has to think about the underlying cause. The HemoSphere/EV1000 with HPI software has a second screen with variables that provide information about the underlying cause of the predicted hypotension.
  Groups: HPI + GDHT treatment

SUMMARY:
The study will investigate whether the use of Goal Directed Hemodynamic Therapy implemented with the HPI algorithm using a treatment algorithm will reduce the incidence of hypotension and improve treatment of hypotension.

DETAILED DESCRIPTION:
The perioperative period is characterized by hemodynamic instability. Intraoperative hypotension (IOH) can be caused by anesthesia drugs, surgical manipulations, hypovolemia or inhibition of the sympathetic nervous system and impairment of baroreflex regulatory mechanisms. In a retrospective analysis performed at the Cleveland Clinic, the risk for acute kidney injury (AKI) and myocardial injury (MI) increased when mean arterial pressure (MAP) was less than 55 mmHg. Further, even short durations of intraoperative hypotension were associated with AKI and MI. Salmasi and coll analyzed whether associations based on relative thresholds were stronger than those based on absolute thresholds regarding blood pressure. They found that there were no clinically important interactions between preoperative blood pressures and the relationship between hypotension and ΜΙ or ΑΚΙ at intraoperative mean arterial blood pressures less than 65 mmHg. Absolute and relative thresholds had comparable ability to discriminate patients with ΜΙ or ΑΚΙ from those without it. The authors concluded that anesthetic management can thus be based on intraoperative pressures without regard to preoperative pressure. In a retrospective cohort study Sun and coll conclude that an increased risk of postoperative stage I AKI occurs when intraoperative MAP was less than 60 mmHg for more than 20 min and less than 55 mmHg for more than 10 min.

Hence it is fundamental for the management of any hemodynamically unstable patient the rapid assessment of the factors that determine the cardiovascular collapse, followed by prompt treatment and, ultimately, reversal of the responsible process. Recently a Hypotension Probability Indicator (HPI) algorithm has been developed from Edwards Lifesciences using continuous invasively-measured arterial waveforms to predict hypotension with high accuracy minutes before blood pressure actually decreases. The HPI algorithm can be integrated with a goal-directed hemodynamic treatment (GDHT) to achieve hemodynamic optimization by increasing global blood ﬂow and prevent organ failure. We developed a treatment protocol implementing HPI with GDHT that can be used in general anesthesia patients to guide clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Planned to receive general anaesthesia > 2h
* Planned to receive an arterial line during surgery
* Aim for MAP of ≥ 65 mmHg during surgery
* Being able to give written informed consent prior to surgery

Exclusion Criteria:

* Aim for MAP other than 65 mmHg at discretion treating physician
* Significant hypotension before surgery defined as a MAP <65
* Right- or left sided cardiac failure (e.g. LVEF<35%)
* Known cardiac shunts (significant)
* Known aortic stenosis (severe)
* Severe cardiac arrhythmias including atrial fibrillation
* Requiring dialysis
* Liver surgery with Pringle maneuver
* Vascular surgery with clamping of the aorta

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We selected adults (age 18 years or older), that underwent surgery lasting for more that 2 hours in which an arterial line was deemed necessary for their hemodynamic monitoring and treatment
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
TWA hypotension (measured with Flotrac sensor) | intraoperative, starting 15 minutes after induction
  Time weighted average spent in hypotension, defined as MAP <65mmHg for ≥1min

SECONDARY OUTCOMES:
Incidence of hypotension (measured with Flotrac sensor) | intraoperative, starting 15 minutes after induction
  Incidence of hypotension, defined as MAP <65mmHg for ≥1min
Time spent in hypotension (measured with Flotrac sensor) | intraoperative, starting 15 minutes after induction
  Time spent in hypotension, in minutes, defined as MAP <65mmHg for ≥1min
Treatment choice (drugs/fluids) | intraoperative, starting 15 minutes after induction
  Medication used to prevent/treat hypotension. A study member is present at the OR to make notes
Treatment dose (drugs/fluids) | intraoperative, starting 15 minutes after induction
  Dose of medication used to prevent/treat hypotension. A study member is present at the OR to make notes
Time to treatment (drugs/fluids) | intraoperative, starting 15 minutes after induction
  time to treatment of hypotension, defined as MAP <65mmHg for ≥1min.
Diagnostic guidance protocol deviations | intraoperative, starting 15 minutes after induction
  Diagnostic guidance protocol deviations, a study member is present at the OR to make notes of any protocol deviations.
Postoperative Morbidity | postoperative, up to 30 days after surgery or until discharge from the hospital
  Incidence of complications: cardiac, pulmonary, renal
Postoperative Creatinine levels | postoperative, up to 30 days after surgery or until discharge from the hospital
  Measurement if creatinine levels postoperatively
Mortality | postoperative, up to 30 days after surgery
  Incidence of mortality 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Sidiropoulou, Principal Investigator — Attikon Hospital
Locations (1):
- Attikon University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
We will share protocol for hemodynamic treatment based on the HPI algorith as well as raw data
Supporting Information: Study Protocol, SAP
Time Frame: We will share data after publication
Access Criteria: individuals who will download/use data must cite location and principal investigator

REFERENCES:
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Background] Sun LY, Wijeysundera DN, Tait GA, Beattie WS. Association of intraoperative hypotension with acute kidney injury after elective noncardiac surgery. Anesthesiology. 2015 Sep;123(3):515-23. doi: 10.1097/ALN.0000000000000765. PMID 26181335